CLINICAL TRIAL: NCT04690231
Title: Apatinib+Ifosfamide and Etoposide (IE) Versus IE Alone for Relapsed or Refractory Osteosarcoma: a Real-world Study in Two Centers in China
Brief Title: Apatinib + Ifosfamide and Etoposide for Relapsed or Refractory Osteosarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 14
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Effect of Drug; Toxicity, Drug; Secondary Resistance
Keywords: osteosarcoma; apatinib; ifosfamide and etoposide; prognosis; toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Osteosarcoma | interventions — apatinib; Ifosfamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib+IE (Experimental)
  Interventions: Drug: Apatinib Mesylate; Drug: ifosfamide and etoposide
- IE (Active Comparator)
  Interventions: Drug: ifosfamide and etoposide

INTERVENTIONS:
Drug: Apatinib Mesylate — apatinib orally daily and ifosfamide 1.8mg/m2/d d1-3, etoposide 100mg/m2/d d1-3
  Other Names: ifosfamide and etoposide
  Arms: Apatinib+IE
Drug: ifosfamide and etoposide — ifosfamide and etoposide

SUMMARY:
Today, using a multi-modal approach consisting of preoperative (neoadjuvant) systemic polychemotherapy followed by local surgical therapy and then postoperative (adjuvant) chemotherapy, long-term, disease-free survival can be achieved in 60- 70% of osteosarcoma patients. However treatment options for osteosarcomas, especially in the setting of metastatic or unresectable disease, are very scarce. Apatinib has been proved to be an effective agent to prolong progression-free survival in advanced osteosarcoma. But after 4-6 months' treatment, secondary resistance always occurred with musculoskeletal lesions' progression or new metastasis.

Nowadays giving therapeutic doses of IE concurrently with anti-angiogenesis tyrosine kinase inhibitors is a conceptually attractive strategy for treating patients with refractory osteosarcoma according to prospective trial of lenvatinib +IE reported by Gaspar et al at 2019 ESMO and 2020 ESMO. Thus This study was designed to review our experience in real world for off-label use and characterize the toxicity profile of concurrent apatinib+IE and IE alone in patients with relapsed or refractory osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of osteosarcoma (confirmed by central pathological review by an expert pathologist from the Peking University People's Hospital)
* objective disease progression within 3 months prior to treatment according to RECIST 1.1
* previously treated with one to two lines of chemotherapy for metastatic disease
* have an adequate performance status (adults:Eastern Cooperative Oncology Group [ECOG] performance status of 0-1;children aged >12 years: a score of ≥60% on the Karnofsky performance scale; children aged ≤12 years a score of ≥60% on the Lansky scale)

Exclusion Criteria:

* a life expectancy of less than 3 months
* patients had to have adequate bone marrow function, normal renal function, normal liver function, and normal pancreatic function
* no other malignant tumors
* no malignant pleural and peritoneal effusion

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
event-free survival | 24 months
  from start treatment to any events/death

SECONDARY OUTCOMES:
progression-free survival | 24 months
  from start treatment to progression/death
overall survival | 24 months
  from start treatment to death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie L, Xu J, Sun X, Tang X, Yan T, Yang R, Guo W. Apatinib for Advanced Osteosarcoma after Failure of Standard Multimodal Therapy: An Open Label Phase II Clinical Trial. Oncologist. 2019 Jul;24(7):e542-e550. doi: 10.1634/theoncologist.2018-0542. Epub 2018 Dec 17. PMID 30559126